CLINICAL TRIAL: NCT04801303
Title: Pilot Trial About the Effects of Calcitriol's Treatment in the Neurological Function and Frataxin's Level in Friedreich's Ataxia Patients
Brief Title: Evaluation of the Effects of Calcitriol's in the Neurological Symptoms of Friedreich's Ataxia Patients
Acronym: CalcitriolFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Berta Alemany (Other)
Collaborators: Institut de Recerca Biomèdica de Lleida (Other); Universitat de Lleida (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor-Investigator, Berta Alemany, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IdIBGI; 2020-001092-32 (EudraCT Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Friedreich Ataxia
Keywords: FA
MeSH Terms: conditions — Friedreich Ataxia | interventions — Calcitriol; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Evaluate the effects of Calcitriol 0.25mcg/24h administered during a year in the neurological symptoms of patients with Friedreich's Ataxia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Friedreich's Ataxia patients (Experimental): Friedreich's Ataxia patients that will receive treatment with Calcitrol 0.25mcg/24h for a year.
  During the clinical trial:
  * The effects of Calcitriol in the neurological symptoms of Friedreich's Ataxia patients will be evaluated before starting the treatment and after a year. The following scales will be used: SARA scale, 9-Hole Peg test, 8 meters walking test, PATA velocity test and Quality of life test with the SF36 questionnaire.
  * The changes in the Frataxin's levels during the treatment with Calcitriol will be measured: before starting the treatment, and after fifteen days, 4 months, 8 months and 12 months of the treatment.
  Interventions: Drug: Calcitriol; Other: Blood analysis for frataxin's level measurement; Diagnostic Test: Blood analysis for hypercalcemia's control

INTERVENTIONS:
Drug: Calcitriol — Administration of Calcitrol 0.25mcg/24h for a year in Friedreich's Ataxia patients (n=20)
  Other Names: Rocaltrol
Other: Blood analysis for frataxin's level measurement — 1. Five blood analysis in Friedreich's Ataxia patients: before starting the treatment, and after fifteen days, 4 months, 8 months and 12 months of the treatment.
  2. To validate the Frataxin's levels measurement, a blood analysis will also be done in two kind of controls for every Friedreich's Ataxia patient, only once at the beginning of the trial.
  The control groups will be composed by:
  * Heterozygous Ataxia's Friedreich controls (a close relative of the patient, either a heterozygous sibling or one of the parents)
  * Age- and gender-matched controls (supposedly non-heterozygous).
Diagnostic Test: Blood analysis for hypercalcemia's control — Five blood analysis in Friedreich's Ataxia patients for monitoring the hypercalcemia risk (with measurement of Calcium, D Vitamin, renal function, albumin, protein, phosphate, sodium and potassium) Before starting the treatment, and after fifteen days, at 4 months, 8 months and 12 months of the treatment.

SUMMARY:
Friedreich's Ataxia (FA) is an autosomal recessive disease the mutation of which leads to a deficiency of a protein called frataxin, which is responsible for the symptoms of the disease. It is assumed that inducing an increase in the production of frataxin could reverse part of the disease's symptoms.

Several treatments with drugs that raise frataxin levels have been tested, but they have either have not given the expected result or have induced intolerable side effects. The IRBLleida (Institut de Recerca Biomèdica de Lleida Fundació Dr. Pifarré) team has shown that calcitriol can increase the production of frataxin up to 2.5 to 3 times, a higher proportion than any of the drugs previously tested. For that reason, the next step in our research would be to check the effects of this drug (Calcitriol 0.25mcg/24h for a year) in patients with FA. On the other hand, calcitriol, the active form of vitamin D, is a drug with a very low rate of adverse effects that has been used for decades. Therefore, it is a drug with a very well established tolerability. The results of the present study, if positive, would lead to the organization of trials at a larger scale, and they would allow the use of an effective treatment for patients with FA.

DETAILED DESCRIPTION:
Friedreich's Ataxia (FA) is a recessive hereditary disease due to GAA (Guanine-Adenosine-Adenosine) triplet repeats in the FXN (Frataxin) gene. This gene codifies for the frataxin protein, the lack of which produces the neurological and cardiac symptoms.

The exact mechanisms why the lack of frataxin produces the disease aren't well understood, but it is known that frataxin is located in the mitochondria. Calcitriol synthesis, a mitochondrial process, could be impaired in FA due the reduction of CYP27B1 (Cytochrome P450, family 27, subfamily B, member 1) and Fdx1.

Because of some studies have shown that Calcitriol (the active form of D Vitamin) could raise the frataxin levels, it could have a beneficial effect in patients with FA.

Description of the trial: to assess the effect of Calcitriol 0.25mcg/24h for a year in the neurological function of FA patients.

Main objective of the trial: to evaluate the effects of Calcitriol in the neurological symptoms of patients with FA.

The second objectives of the trial are:

1. To evaluate the safety and the risk of hypercalcemia with the treatment with low dosis of Calcitriol (0.25mcg of Calcitriol every 24h) in patients with FA.
2. To measure de change in the Frataxin's levels during the treatment with Calcitriol.
3. To evaluate the effects of Calcitriol in the daily life activities and the life quality of the patients with FA.

Sample size: The number of participants needed to compleat the trial is 20. Duration: The duration of the trial is one year

Procedure:

* Before taking part in the study, it will be ensured that participants fulfill all the inclusion criteria with a detailed questionnaire.
* During the clinical trial the following test will be done: 4 electrocardiogram, 5 blood analysis to control de risk of hypercalcemia and to measure the frataxin's levels, and 3 full neurological examinations.

Post trial treatment details:

The patients who wish to continue with the treatment will be allowed to do so, at least until the results of the comparison of the basal neurological evaluation with the second and the final neurological evaluation are obtained.

If the results are positive, the treatment will be continued with regular blood tests controls.

If the results don't demonstrate a statistically significant effect, the treatment will be interrupted in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Friedreich's Ataxia and confirmed genetic diagnosis with:

  * Two pathological GAA triplet repeats in the gen FXN
  * One pathological GAA triplet repeat and one point mutation in the gen FXN
* Patients between 16 and 65 years of age.
* To keep the walking ability, although an external aid is needed.
* Women with confirmed genetic diagnosis must use an effective contraceptive method during the trial.

Exclusion Criteria:

* Any neurological or other kind of disease that could interfere in the trial according to the investigator judgement.
* Severe visual loss.
* Severe auditory loss.
* Cognitive decline*.

  * Dementia or affective-cognitive cerebellar syndrome.
* Serious psychiatric illness during the six previous months of the trial inclusion.
* Substance abuse during the six previous months of the trial inclusion.
* Severe drug allergy.
* Cardiac disease:

  * Ejection fraction <40% [N: 50-70%]
  * Heart failure > 2 from NYHA (New York Heart Association) criteria.
  * Significant valvular heart disease.
  * Symptomatic coronary artery disease.
  * Cardiac arrhythmia with hemodynamic compromise (atrial fibrillation).
* Prolonged immobilisation
* Use of research drugs during the 30 previous days of the trial inclusion.
* Concomitant treatment with digoxin, thiazide diuretics, cholestyramine, corticoids, laxatives with magnesium, barbiturates and antiepileptic drugs. Use of Calcium or Vitamin D drugs during the 30 previous days of the trial inclusion.
* Legally or mentally incapacitated person.
* In women:

  * Positive pregnancy test.
  * Maternal breastfeeding.
* Blood test alteration:

  * Hypercalcemia.
  * Elevated creatinine.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in the SARA scale (Scale for the Assessment and Rating of Ataxia) in FA patients after a one-year treatment with Calcitriol. | At the beginning, and at the 6th and 12th month (one year) after the beginning of the trial.
  SARA is a scale which assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
  The eight categories have an accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
  When completing the outcome measure each category is assessed and scored accordingly. Scores for the eight items range as follows:
  * Gait (0-8 points),
  * Stance (0-6 points),
  * Sitting (0-4 points)
  * Speech disturbance (0-6 points)
  * Finger chase (0-4 points)
  * Nose-finger test (0-4 points)
  * Fast alternating hand movement (0-4 points)
  * Heel-shin slide (0-4 points) Once each of the 8 categories have been assessed, the total is calculated to determine the severity of ataxia.
Changes in the 9-Hole Peg test in FA patients after a one-year treatment with Calcitriol. | At the beginning, and at the 6th and 12th month (one year) after the beginning of the trial.
  The 9-Hole Peg test is a quantitative assessment used to measure fingir dexterity.
  It is administered by asking the participant to take de pegs from a container, one by one, and place them into the holes on the boward, as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. The board should be placed at the client's midline, with the container holding the pegs oriented towards the hand being tested.
  Only the hand being evaluated should perform the test. Hand not being evaluated is permitted to hold the edge of the board in order to provide stability. Both hands will be assessed.
  Scores are recorded in seconds and are based on the time taken to complete the test activity, scoring better when less seconds are required to complete de test. Stopwatch should be started from the moment the participant touches the first peg until the moment the last peg hits the container.
Changes in the 8 meters walking test in FA patients after one year treatment with Calcitriol. | At the beginning, and at the 6th and 12th month (one year) after the beginning of the trial.
  The 8 meters waking test is used to asses walking speed in over a short distance of 8 meters. It is administered by asking the participant to walk through an 8 meteres lenght stright line as faster as posible.
  Scores are recorded in seconds and are based on the time taken to complete the test activity, scoring better when less seconds are required to complete de test.
  Stopwatch should be started from the moment the participant starts to walk until he reaches the final of the stright line.
Changes in the PATA rate test in FA patients after one year treatment with Calcitriol. | At the beginning, and at the 6th and 12th month (one year) after the beginning of the trial.
  PATA Rate Task is a quantitative test used to measure the severity of dysarthria.
  Participants are invited to repeat the syllables "PA-TA" as quickly as possible during a 10 seconds interval. They will do the same test twice, being the final score the average of the two attempts.
  The score consists in the number of correct repetition of both syllables, scoring better when they are able to say more correct repetitions of the syllables.
Changes in Barthel index for Activities of Daily Living in FA patients after one year treatment with Calcitriol. | At the beginning, and at the 12th month (one year) after the beginning of the trial.
  Barthel index is an objective, standardized tool for measuring functional status. The individual is scored in a number of areas depending upon independence of performance.
  The ten variables measured in the Barthel scale are:
  * Presence or absence of fecal incontinence
  * Presence or absence of urinary incontinence
  * Help needed with grooming
  * Help needed with toilet use
  * Help needed with feeding
  * Help needed with transfers (e.g. from chair to bed)
  * Help needed with walking
  * Help needed with dressing
  * Help needed with climbing stairs
  * Help needed with bathing The total score range from 0, that is equivalent to complete dependence, to 100, that is equivalent to complete independence.
Changes in SF36 questionnaire in FA patients after one year treatment with Calcitriol. | At the beginning, and at the 12th month (one year) after the beginning of the trial.
  The SF-36 questionnaire is a qualitiy life teast to assess the quality of life. It contains 36 questions that address different aspects related to the daily life of the person who fills in the questionnaire.
  These questions are grouped and measured in 8 sections that are evaluated independently. The 8 dimensions included in each section are:
  * Physical functioning.
  * Limitations due to physical problems.
  * Body pain.
  * Social functioning.
  * Mental health.
  * Limitations due to emotional problems.
  * Vitality, energy or fatigue.
  * General perception of health. The questionnaire questions ask for answers related to the previous month. The scores for each of the 8 dimensions of the SF-36 range between the values 0 and 100, with 100 being a result that indicates optimal health and 0 would reflect a very poor state of health.
Changes in Frataxin's levels during Calcitriol treatment.. | At the beginning, and at the 15th day, 4th month, 8th month and 12th month after the beginning of the trial.
  In FA patients will be done blood analysis to monitor de Frataxin's levels.
  To validate the Frataxin's levels measurement a blood analysis will also be done in two kind of controls for every FA patient:
  * One heterozygous FA control (a close relative of the patient, either an heterozygous sibling or one of the parents).
  * One age- and gender-matched control, supposedly non-heterozygous. The controls should not have any neurological or related with Calcium metabolism disease, or should not be under treatment with Calcium or D Vitamin.

SECONDARY OUTCOMES:
Assessing the Calcitriol treatment's side effects with an hypercalcemia symptoms' questionnaire. | At the 15th day, 4th month, 8th month and 12th month after the beginning of the trial.
  In the hypercalcemia symptom's questionnaire the following items are asked and answered with a "yes" or "no" answer:
  * The development or presence of headache.
  * The development or presence of nausea.
  * The development or presence of abdominal pain.
  * The development or presence of polyuria.
  * The development or presence of a skin rash. When one or more questions are answered with a "Yes" means that may exist a side effect due the Calcitriol treament.
Assessing the Calcitriol treatment's hypercalcemia risk with an Electrocardiogram (ECG). | At the beginning, and at the 15th day, 4th month, 8th month and 12th month after the beginning of the trial.
  The ECG is an electrical record of the function of the heart. It is used a 12-lead ECG, placed in the chest and arms and leds, that detect the small electrical changes that are a consequence of cardíac muscle depolarization followed by repolarization during each cardíac cycle (heartbeat).
  It is recorded the heartrate, the P wave lenght, the QRS complex lenght and form and the QT interval. The shortening of the QT interval, measured in seconds, indicates a electrocardiographyc alteration due an hypercalcemia.
Assessing the treatment's hypercalcemia risk with a blood test. | At the beginning, and at the 15th day, 4th month, 8th month and 12th month after the beginning of the trial.
  The blood test is a laboratory analysis performed on a blood sample that usually is extracted from a vein in the arm using a hypodermic needle. Different measures can be obtained from a single blood test. In order to assess de hypercalcemia risk there are analyzed the levels of Calcium, 1-25-dihydroxi-Colecalciferol, Phosphorus, Albumin, Proteins, Creatinine, Urea, Sodium and Potassium.
  The measurament that indicates an hypercalcemia risk are:
  * Calcium levels > 10.2 mg/dl. The Albumin and Proteins analysis is needed for the measurement of Calcium level.
  * 1-25-dihydroxi-Colecalciferol levels > 100 ng/ml
  * Phosphorus levels > 4.5 mg/dl
  The hypercalcemia risk is higher when coexists a renal insufficiency. The measuramenst that indicates a renal insufficiency are:
  * Creatinine > 1.2 mg/dl
  * Urea > 48.5 mg/dl
  * Sodium > 145 mEq/L
  * Potassium > 5.1 mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Berta Alemany Perna, Principal Investigator — Hospital Universitari Josep Trueta/Hospital Santa Caterina, Girona/Salt, Spain
Locations (1):
- Hospital Santa Caterina/Parc Martí i Julià, Salt, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Britti E, Delaspre F, Sanz-Alcazar A, Medina-Carbonero M, Llovera M, Purroy R, Mincheva-Tasheva S, Tamarit J, Ros J. Calcitriol increases frataxin levels and restores mitochondrial function in cell models of Friedreich Ataxia. Biochem J. 2021 Jan 15;478(1):1-20. doi: 10.1042/BCJ20200331. PMID 33305808

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04801303/Prot_SAP_000.pdf
  • Informed Consent Form: Healthy control informed consent form (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT04801303/ICF_001.pdf
  • Informed Consent Form: Healthy control informed consent form (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT04801303/ICF_002.pdf